CLINICAL TRIAL: NCT03773250
Title: A FAMILY Program for Childhood Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201603121RIND
Record Dates: First submitted 2018-10-23; First posted 2018-12-12 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): Children and families in the intervention group will received the FAMILY program developed according to evidence-based guidelines.The intervention content regarding healthy sleep will emphasize the importance of having a consistent sleep schedule, establishing a regular bedtime routine, and creating an environment only for sleeping. The physical activity content will emphasize at least 60 minutes/day of moderate-to-vigorous intensity physical activity, reduction of sedentary behavior, and screen time limited to 2 hours/day. The nutrition content will emphasis the replacement of sugar-sweetened beverages, increased fruit and vegetable as well as water intake, consumption of regular meals, and reduction of discretionary food groups.
  Interventions: Behavioral: Behavioral intervention
- Control (Other): An active placebo control intervention was designed which did not apply evidence-based lifestyle recommendations effective in weight loss and focused on vegetable education.
  Interventions: Behavioral: Behavioral intervention

INTERVENTIONS:
Behavioral: Behavioral intervention — The intervention has an intensive phase and a maintenance phase.

SUMMARY:
Childhood overweight and obesity is a health problem with lifelong implications related to diabetes, hypertension, cardiovascular disease, psychological disorders as well as other chronic conditions.

DETAILED DESCRIPTION:
In Taiwan, the nationwide prevalence of overweight and obesity among school-age children aged 7 to 11 years has also increased over the past years. Sleep and weight are intricately related. School-age children requires at least 10 hours of sleep per night but children in Asian countries are on average obtaining shorter sleep than children in Caucasian countries.

ELIGIBILITY:
Inclusion Criteria:

* Children with overweight and obesity

Exclusion Criteria:

* Children with any other chronic or acute medical conditions

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Child BMI-for-age z-score | Change from baseline to 12 months post intervention
  Child BMI-for-age z-score will be computed based on the World Health Organization growth reference data for 5-19 years.

SECONDARY OUTCOMES:
Child BMI | Change from baseline to 12 months post intervention
  Child BMI will be calculated based on child weight and height.
Child percent body fat | Change from baseline to 12 months post intervention
  Percent body fat will be estimated according to the skinfold thickness equations.
child sleep duration and sleep efficiency | Change from baseline to 12 months post intervention
  Actigraphy-derived daily sleep duration and nocturnal sleep efficiency
Parental sleep quality | Change from baseline to 12 months post intervention
  Pittsburgh Sleep Quality Index total scores

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Tsai, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No